CLINICAL TRIAL: NCT02249624
Title: The Utility of MRI Scoring to Predict Neurodevelopmental Outcomes in Survivors
Brief Title: The Utility of MRI Scoring to Predict Neurodevelopmental Outcomes in Survivors of Twin-to-Twin Transfusion Syndrome
Status: Completed | Type: Observational
Sponsor: Catherine Cibulskis, MD (Other)
Collaborators: St. Louis University (Other)
Responsible Party: Sponsor-Investigator, Catherine Cibulskis, MD, Assistant Professor of Pediatrics, St. Louis University
Organization: St. Louis University (Other)
Other Study IDs: 23854
Record Dates: First submitted 2014-09-15; First posted 2014-09-25 (Estimated); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Fetofetal Transfusion
Keywords: Twin to twin transfusion syndrome; Developmental disabilities; Magnetic resonance imaging
MeSH Terms: conditions — Fetofetal Transfusion; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survivors of TTTS: Infants who have survived TTTS to hospital discharge, have an MRI at term, and return for nursery follow-up clinic.

SUMMARY:
Twins who share a placenta but have two separate sacs of amniotic fluid (monochorionic-diamniotic) are at risk of developing twin-to-twin transfusion syndrome (TTTS). TTTS results from anastomoses in the placenta that lead to unequal sharing of blood, causing abnormal blood flow to the twins. The donor twin may have low fluid levels, poor growth, and anemia. The recipient twin can have high fluid levels, high red blood cell counts, heart failure, and hydrops. Having TTTS, especially if there is demise of one twin or if disease is severe enough to warrant laser photocoagulation of the anastomotic sites, puts the surviving fetuses at risk for brain injury due to hypoxia, ischemia, or reperfusion injuries. Magnetic Resonance Imaging (MRI) is superior to ultrasound at detecting subtle cerebral injuries. An MRI scoring scale has been developed for use in very low birth weight infants that has been shown to correlate with neurodevelopmental outcomes, but it has not been tested in this patient population.

Our center's guidelines recommend fetal MRI prior to intervention, at 32 weeks gestational age, and on the infants at term corrected gestational age. Infants who were treated for TTTS in utero are seen in Nursery Follow-up Clinic at 4 months of age, 8 months of age, and for Bayley Scales evaluations at 15-18 months of age and at 2-3 years of age.

The purpose of this study is to correlate brain MRI score with neurodevelopmental outcomes in survivors of TTTS that have either required fetal surgical intervention or had demise of their cotwin. The investigators predict that more severe white and gray matter injury as determined by the Woodward/Inder grading scale will be positively associated with worse neurodevelopmental outcomes.

DETAILED DESCRIPTION:
All mothers with a pregnancy affected by twin-to-twin transfusion syndrome (TTTS) who are referred to the St. Louis Fetal Care Institute (FCI) will be evaluated for enrollment over a two year period. The women who have severe findings that indicate a need for fetal intervention or who had demise of one fetus due to TTTS will be approached at FCI to discuss the study. Once the baby(ies) is/are born, written consent for the infant's participation will be obtained.

FCI and Cardinal Glennon Children's Medical Center have an established protocol for TTTS. Fetuses affected by TTTS under fetal MRI and echocardiogram at the time of diagnosis (if time permits before intervention) and again at 32 weeks of gestation. The infants receive a postnatal MRI at term corrected gestational age (>37 weeks of gestation). This may be done as an inpatient if they are still hospitalized at Cardinal Glennon, or as an outpatient if their birth hospitalization was at a different hospital, or if they are discharged to home prior to 37 weeks of age. They also receive a postnatal echocardiogram, which may be done during the birth hospitalization, or at the time of their outpatient MRI appointment. All of the infants are followed at 4-6 months of age for physical therapy evaluation, and if there are concerns, they return 4 months later for a repeat physical therapy evaluation. Bayley Scales of Infant Development (BSID-III) evaluations are performed by a child psychologist at 15-18 months corrected age, and again between 2-3 years of age. At any time in this process, if there are concerns about developmental progress, home therapy services are prescribed to help improve outcomes.

This protocol of evaluations results in a total of 3-5 follow-up appointments for each infant after initial hospital discharge, and are all standard of care at the investigators hospital.

MRI provides more detailed information than ultrasound in diagnosing hypoxic ischemic brain damage both prenatally and postnatally (1,2). Ultrasound has low sensitivity to detect non-hemorrhagic brain injuries, and studies have shown that only 14-27% of infants with cerebral injury on MRI had any abnormalities seen on head ultrasound(3,4).

Studies in premature infants have shown a correlation between MRI findings at term corrected age and neurodevelopmental outcomes. A grading scale has been proposed by Woodward and Inder to assess the degree of white and gray matter injury on MRI(5-7). After multivariate adjustment, this scale showed that increasing severity of white matter abnormalities was associated with increased risks of severe motor delay and cerebral palsy (5). The presence of any white matter abnormalities was found to be more sensitive at identifying children who had neurodevelopmental impairments than ultrasound findings of intraventricular hemorrhage or periventricular leukomalacia(5). Furthermore, most children with a normal or only mildly abnormal MRI were free of severe impairments at 2 years of age(5).

If infants at highest risk of neurodevelopmental delays could be identified earlier and more accurately, these infants could be monitored more closely and earlier interventions could be administered. This would potentially result in better long-term neurodevelopmental outcomes for these high-risk children. However, there is currently no correlative data between MRI findings and long-term neurodevelopmental outcomes in the survivors of TTTS.

ELIGIBILITY:
Inclusion Criteria:

* Infants who suffered from TTTS in utero that either required fetal laser photocoagulation or had death of their cotwin
* Born after implementation of our TTTS protocol in September 2013
* Complete postnatal MRI and follow-up at Cardinal Glennon Children's Medical Center, or at an outside hospital and release medical information to the study

Exclusion Criteria:

* Infants who did not have TTTS, or not severe enough to warrant fetal intervention or demise of the cotwin
* Infants who do not complete their follow-up per protocol

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pregnancies affected by TTTS will be identified through referrals from the St. Louis Fetal Care Institute. Surviving infants of those pregnancies that required fetal laser surgery, or had death of the cotwin, will be approached for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-09; Primary Completion 2020-09-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Composite outcome of neurodevelopmental impairment - final | 3 years of age
  Defined by mental, language, or physical developmental index < 2 standard deviations from the mean on the Bayley Scales of Infant Development III, neurosensory impairment (hearing loss requiring aids or blindness), or the diagnosis of cerebral palsy.

SECONDARY OUTCOMES:
Developmental delay - 4 months | 4 months of age
  Defined by delays of >1 month on physical therapy evaluation at 4 months of age
Developmental delay - 8 months | 8 months of age
  Defined by delays of >1 month on physical therapy evaluation at 8 months of age
Neurodevelopmental impairment - 15 months | 15 months of age
  Defined by mental, language, or physical developmental index < 2 standard deviations from the mean on the Bayley Scales of Infant Development III
MRI results | Term gestational age
  Score on MRI, and pattern of MRI findings on donor and recipient twins when they reach term corrected gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cibulskis, MD, Principal Investigator — St. Louis University
Locations (1):
- Cardinal Glennon Children's Medical Center, St Louis, Missouri, United States

REFERENCES:
- [Background] Simonazzi G, Segata M, Ghi T, Sandri F, Ancora G, Bernardi B, Tani G, Rizzo N, Santini D, Bonasoni P, Pilu G. Accurate neurosonographic prediction of brain injury in the surviving fetus after the death of a monochorionic cotwin. Ultrasound Obstet Gynecol. 2006 May;27(5):517-21. doi: 10.1002/uog.2701. PMID 16586472
- [Background] Righini A, Kustermann A, Parazzini C, Fogliani R, Ceriani F, Triulzi F. Diffusion-weighted magnetic resonance imaging of acute hypoxic-ischemic cerebral lesions in the survivor of a monochorionic twin pregnancy: case report. Ultrasound Obstet Gynecol. 2007 Apr;29(4):453-6. doi: 10.1002/uog.3967. PMID 17390325
- [Background] Merhar SL, Kline-Fath BM, Meinzen-Derr J, Schibler KR, Leach JL. Fetal and postnatal brain MRI in premature infants with twin-twin transfusion syndrome. J Perinatol. 2013 Feb;33(2):112-8. doi: 10.1038/jp.2012.87. Epub 2012 Jun 28. PMID 22743408
- [Background] Inder TE, Anderson NJ, Spencer C, Wells S, Volpe JJ. White matter injury in the premature infant: a comparison between serial cranial sonographic and MR findings at term. AJNR Am J Neuroradiol. 2003 May;24(5):805-9. PMID 12748075
- [Background] Woodward LJ, Anderson PJ, Austin NC, Howard K, Inder TE. Neonatal MRI to predict neurodevelopmental outcomes in preterm infants. N Engl J Med. 2006 Aug 17;355(7):685-94. doi: 10.1056/NEJMoa053792. PMID 16914704
- [Background] Inder TE, Wells SJ, Mogridge NB, Spencer C, Volpe JJ. Defining the nature of the cerebral abnormalities in the premature infant: a qualitative magnetic resonance imaging study. J Pediatr. 2003 Aug;143(2):171-9. doi: 10.1067/S0022-3476(03)00357-3. PMID 12970628
- [Background] Woodward LJ, Mogridge N, Wells SW, Inder TE. Can neurobehavioral examination predict the presence of cerebral injury in the very low birth weight infant? J Dev Behav Pediatr. 2004 Oct;25(5):326-34. doi: 10.1097/00004703-200410000-00004. PMID 15502549